CLINICAL TRIAL: NCT01922011
Title: A Multicenter, Randomized, Double-Blinded Comparative Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Daptomycin Versus Active Comparator in Pediatric Subjects With Acute Hematogenous Osteomyelitis Due to Gram-Positive Organisms
Brief Title: Safety and Efficacy Study of Daptomycin Compared to Active Comparator in Pediatric Participants With Acute Hematogenous Osteomyelitis (AHO) (MK-3009-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3009-006; DAP-PEDOST-11-03 (Other: Cubist Pharmaceuticals, Inc. Protocol Number); 2013-000864-28 (EudraCT Number)
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Acute Hematogenous Osteomyelitis
MeSH Terms: interventions — Daptomycin; Vancomycin; Nafcillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daptomycin (Experimental): Intravenous (IV) daptomycin was dosed as follows: age 12 years to <18 years (7 mg/kg); age 7 years to < 12 years (9 mg/kg); age 24 months to <7 years (12 mg/kg); age 12 months to <24 months (12 mg/kg). Drug was infused over 60 minutes ± 10 minutes once daily followed by up to 3 dummy infusions every 6 hours (q6h) infused over 60 (± 10) min to maintain the blind.
  Interventions: Drug: Daptomycin
- Vancomycin or Nafcillin (Active Comparator): IV vancomycin (or equivalent), 10 to 15 mg/kg, was infused over 60 (± 10) minutes q6h (± 1 hour) or IV nafcillin (or β-lactam equivalent) at 100-200 mg/kg/day, in divided doses was infused over 60 (± 10) min q6h (± 1 hour)
  Interventions: Drug: Vancomycin (or equivalent); Drug: Nafcillin (or equivalent)

INTERVENTIONS:
Drug: Daptomycin — IV daptomycin Infusion A in 12 to <18 years old (7 mg/kg); in 7 to < 12 year olds (9 mg/kg); in 24 months to <7 year olds (12 mg/kg); in 12 to <24 month olds (12 mg/kg). Infused over 60 minutes ± 10 minutes once daily followed by up to 3 dummy infusions every 6 hours (q6h) infused over 60 (± 10) min to maintain the blind.
  Arms: Daptomycin
Drug: Vancomycin (or equivalent) — IV vancomycin (or equivalent) (Infusions A,B,C,D), 10 to 15 mg/kg, infused over 60 (± 10) minutes q6h (± 1 hour)
  Arms: Vancomycin or Nafcillin
Drug: Nafcillin (or equivalent) — IV nafcillin (or β-lactam equivalent) (Infusions A,B,C,D) at 100-200 mg/kg/day, in divided doses infused over 60 (± 10) min q6h (± 1 hour)
  Arms: Vancomycin or Nafcillin

SUMMARY:
The purpose of the study is to determine whether daptomycin is effective and safe in the treatment of pediatric participants with AHO when compared to vancomycin (or equivalent) or nafcillin (or β-lactam equivalent). The primary hypothesis is that daptomycin is non-inferior compared with vancomycin (or equivalent) or nafcillin (or β-lactam equivalent) with respect to improvement in Pain, Inflammation, and Limb Function on or before study Day 5.

DETAILED DESCRIPTION:
Acute hematogenous osteomyelitis is a common problem in the pediatric population, affecting approximately 5/10,000 children each year and accounting for approximately 1% of all pediatric hospitalizations. In children, osteomyelitis arises from bacteremic seeding of the bone metaphysis.

Daptomycin, is a cyclic lipopeptide antibacterial active against most clinically significant gram-positive pathogens including drug-resistant strains such as Methicillin Resistant Staphylococcus (S.) aureus (MRSA) and Methicillin Susceptible S. aureus (MSSA). Daptomycin has proven clinical efficacy in adults in the treatment of complicated skin and skin structure infections (cSSSI) caused by aerobic gram-positive pathogens and the treatment of S. aureus bloodstream infections (bacteremia; SAB), including those complicated by right-sided infective endocarditis, caused by MSSA and MRSA. Although not indicated for osteomyelitis, daptomycin has been successfully used to treat osteoarticular infections in adults and children as salvage therapy and at medical centers with increasingly high rates of vancomycin resistant organisms.

In addition, more comparative clinical trials are needed in pediatric AHO to better elucidate the optimal treatment regimen and clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Obtain Informed Consent;
* Be 1 year to < 18 years old; a stepwise approach will be implemented to gate enrollment as follows: enrollment will begin with children aged 2-17 years; after an external Drug Safety Monitoring Board (DSMB) review, enrollment will be broadened to 1-17 years.
* Have diagnosis of suspected or confirmed AHO warranting IV antibacterial therapy as inpatient, based on clinical, imaging and/or microbiological evidence as outlined below:

I. Clinical evidence of fever accompanied by symptoms on the affected limb that include but it is not limited to pain, tenderness on palpation, inflammation, warmth, swelling, difficulty bearing weight, motion restriction, loss of function

II. Radiologic imaging (magnetic resonance imaging [MRI], bone scan, x-ray, or computed tomography [CT] scan) consistent with osteomyelitis OR Microbiological evidence (gram stain, culture or polymerase chain reaction (PCR)) from a bone biopsy or bone aspirate (if available), or blood

III. Laboratory evidence: C-reactive protein (CRP) elevated, Erythrocyte sedimentation rate (ESR) elevated, leukocytosis or leukopenia, immature neutrophils

•Confirmed (I, II, and III) OR suspected (I and III) that must be confirmed post-randomization

Participants will not be allowed into the study if they:

* Have documented history of any hypersensitivity or allergic reaction to daptomycin
* Have septic arthritis only (without AHO)
* Have acute hematogenous osteomyelitis that is located in the spine
* Have chronic osteomyelitis (i.e. symptoms of osteomyelitis > 21 days) or osteomyelitis with complications requiring non-routine surgical treatment (i.e. sequestration).
* Have major trauma, penetrating trauma (including a puncture wound of the foot), postoperative osteomyelitis, foreign body in or adjacent to affected bone or joint, or other iatrogenic bone or joint infections present at the site of infection
* Have acute hematogenous osteomyelitis due to a proven gram-negative organism
* Have transient tenosynovitis, juvenile rheumatoid arthritis (JRA), reactive arthritis, bony tumors, and other osteoarticular diseases suspected to be due to a nonbacterial (eg, fungal or mycobacterial) etiology
* Receive more than 24 hours of effective intravenous antibacterial therapy for osteomyelitis within 96 hours before randomization unless microbiological or clinical failure is documented
* Require any potentially effective concomitant systemic antibacterial therapy for gram-positive infections
* Have history of seizures (except febrile seizure of childhood)
* Have peripheral neuropathy
* Have history of rhabdomyolysis (with the exception of muscle injury due to trauma)
* Have Sickle cell anemia
* Cannot be assessed clinically during the study
* Have any condition (eg, cystic fibrosis, current septic shock) that would make the subject, in the opinion of the Investigator, unsuitable for the study
* Have significant reduced creatinine clearance (CrCl) < 50 mL/min/1.73 m2
* Have evidence of significant hepatic, hematologic, or immunologic dysfunction
* Have Creatine kinase (CK) elevation ≥ 10 × ULN (upper limit of normal) without symptoms or ≥ 5 × ULN with symptoms
* If female, must not be pregnant or nursing and if required by age and life style take appropriate measures to not get pregnant during the study.
* Have participated in any study involving administration of an investigational agent or device or daptomycin within 30 days
* Are unable or unwilling to adhere to the study-specified procedures and restrictions
* Has suspected or confirmed pneumonia, empyema, meningitis, or endocarditis.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Bradley JS, Arrieta AC, Digtyar VA, Popejoy MW, Grandhi A, Bokesch P, Hershberger E, Dorr MB, Tan CM, Murata Y, Wolf DJ, Bensaci M. Daptomycin for Pediatric Gram-Positive Acute Hematogenous Osteomyelitis. Pediatr Infect Dis J. 2020 Sep;39(9):814-823. doi: 10.1097/INF.0000000000002790. PMID 32639465

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin: Intravenous (IV) daptomycin 7, 9, or 12 mg/kg once daily and ≤3 dummy infusions daily
- Vancomycin or Nafcillin: IV vancomycin (or equivalent), 10 to 15 mg/kg every six hours (q6h), or IV nafcillin (or β-lactam equivalent) 100-200 mg/kg/day, in divided doses q6h.
Period: Overall Study
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Started | 75 (Randomized participants) | 74 (Randomized participants)
Treated | 73 (Treated Participants) | 73 (Treated Participants)
Treatment Actually Received | 74 (One participant intended for treatment with Vancomycin or Nafcillin was treated with Daptomycin) | 72 (One participant intended for treatment with Vancomycin or Nafcillin was treated with Daptomycin)
Completed | 69 | 69
Not Completed | 6 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Parent/Guardian Decision | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Missed Test-of-Cure Visit | 0 | 2
Not completed — Not Treated | 1 | 0
Not completed — Lack of willing home health agency | 1 | 0
Not completed — Randomized in error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Daptomycin: IV daptomycin 7, 9, or 12 mg/kg once daily and ≤3 dummy infusions daily
- Vancomycin or Nafcillin: IV vancomycin (or equivalent), 10 to 15 mg/kg q6h, or IV nafcillin (or β-lactam equivalent) 100-200 mg/kg/day, in divided doses q6h.
- Total: Total of all reporting groups
Arm/Group | Daptomycin | Vancomycin or Nafcillin | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.1 (4.4) | 9.2 (4.1) | 9.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 56
  Male | 44 | 49 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Improvement in the 3 General Categories of Pain, Inflammation, and Limb Function Based on the Investigator's Overall Assessment of Severity of Each of the Symptom Categories.
Description: Clinical improvement was based on the Investigator's overall assessment of severity of each of the 3 general symptom categories of Pain, Inflammation, and Limb Function. Based on this evaluation, a participant was considered to have met criteria for clinical improvement according to the following definition: If 3 general categories are present at baseline: at least a 1-point improvement (i.e. severe to moderate, moderate to mild, mild to absent) in at least 2 of the general categories and no worsening in the other. If 2 general categories are present at baseline: at least a 2-point improvement (i.e. severe to mild, moderate to absent) in at least 1 of the general categories and no worsening or new findings in the others OR at least a 1-point improvement in both and no new findings in the other. If 1 general category is present at baseline: at least a 2-point improvement (i.e., severe to mild, moderate to absent) in that category and no new findings in the others.
Time Frame: Up to study Day 5
Population: All randomized participants who received any amount of IV study drug and who had a confirmed or suspected diagnosis of AHO, excluding those with confirmed culture of a gram-negative organism from any baseline specimen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 71 | 70
Percentage of participants | 77.5 [67.7 to 87.2] | 82.9 [74.0 to 91.7]
Statistical Analysis 1: Comparison: Daptomycin vs Vancomycin or Nafcillin; 95% confidence interval of the common difference was based on stratified Newcombe confidence interval (CI) with minimum risk weights, with age cohort as the stratification factor; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower bound of the 2-sided 95% CI is greater than -15%; p = 0.421, Wald; Common Difference = -6.1, 95% CI 2-sided [-19.4 to 7.4] — Daptomycin - Comparator

2. Secondary Outcome: Percentage of Participants With Clinical Improvement Measured as a Composite End Point of Pain, Inflammation, Limb Function, Body Temperature, and C-reactive Protein at End-of IV (EOIV) Therapy Visit.
Description: A participant had a favorable outcome in this composite endpoint if all 3 of the following criteria were met: Clinical improvement in the general symptom categories of Pain, Inflammation, and Limb Function on or before Study Day 5; Body temperature ≤ 38°C (100.4°F) over the preceding 24 hours; and C-reactive Protein (CRP) decreased from baseline for participants who had a baseline CRP >ULN (upper limit of normal)) or remain <=ULN for participants who had a baseline <=ULN on or before Study Day 5. The EOIV visit is within 24 hours after the last dose of IV study drug and before switch to optional open label (PO) therapy, if applicable.
Time Frame: Up to study Day 5
Population: All randomized participants who received any amount of IV study drug and who had a confirmed diagnosis of AHO (Categories I, II and III), excluding participants with confirmed culture of a gram-negative organism from any baseline specimen and who did not have all clinical assessments performed at the time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 69 | 68
Percentage of participants | 71.0 [60.3 to 81.7] | 76.5 [66.4 to 86.6]
Statistical Analysis 1: Comparison: Daptomycin vs Vancomycin or Nafcillin; Test type: Superiority or Other; p = 0.467, Wald; Common difference = -7.1, 95% CI 2-sided [-21.6 to 7.9] — 95% confidence interval of the common difference ( Daptomycin minus Vancomycin or Nafcillin) is based on stratified Newcombe confidence interval (CI) with minimum risk weights, with age cohort as the stratification factor

3. Secondary Outcome: Percentage of Participants With a Favorable Clinical Outcome
Description: Favorable clinical outcomes are clinical recovery and clinical cure. Clinical cure is defined as resolution of all acute symptoms of AHO or improvement to such an extent that no further intravenous antibacterial therapy is required. Clinical recovery is defined as clinical improvement in the composite end point three general categories of Pain, Inflammation, and Limb Function on or before Study Day 5, and no development of new symptoms of AHO; body temperature ≤ 38°C (100.4°F) for 24 hours; no new or additional bone or joint infection (e.g., abscess, spreading to other osseous or articular locations) such that no further antibacterial therapy or surgery are required; no hematogenous metastatic infection (e.g., abscess in liver, spleen, lung; other bones) or bacteremia.. The End of Therapy (EOT) visit is within 48 hours of last dose of PO therapy.
Time Frame: Baseline (within 48 hours prior to first dose of IV study drug) - and up to Test of Cure (21-35 days after last dose of IV study drug) (up to Day 77)
Population: All randomized participants who received any amount of IV study drug and who had a confirmed diagnosis of AHO (Categories I, II and III), excluding participants with confirmed culture of a gram-negative organism from any baseline specimen
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 71 | 70
Percentage of participants
  At End of IV (EOIV) Therapy (n= 71,69) | 85.9 [77.8 to 94.0] | 91.3 [84.7 to 98.0]
  At End of Therapy (EOT) (n= 71,69) | 83.1 [74.4 to 91.8] | 89.9 [82.7 to 97.0]
  At Test Of Cure (TOC) (n= 71,70) | 81.7 [72.7 to 90.7] | 87.1 [79.3 to 95.0]
Statistical Analysis 1: Comparison: Daptomycin vs Vancomycin or Nafcillin; At EOIV visit; Test type: Superiority or Other; p = 0.313, Wald; Common difference = -6.2, 95% CI 2-sided [-17.5 to 5.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Daptomycin vs Vancomycin or Nafcillin; At EOT visit; Test type: Superiority or Other; p = 0.239, Wald; Common difference = -7.9, 95% CI 2-sided [-19.8 to 4.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Daptomycin vs Vancomycin or Nafcillin; At TOC visit; Test type: Superiority or Other; p = 0.370, Wald; Common difference = -6.7, 95% CI 2-sided [-19.1 to 5.8] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With a Clinical Cure Categorized by Baseline Pathogen at Test of Cure
Description: At Test Of Cure (TOC) clinical cure is defined as resolution of all acute symptoms of AHO or improvement to such an extent that no further antibacterial therapy is required. Favorable microbiological outcomes are either eradication where the source specimen demonstrated absence of the original baseline pathogen; or presumed eradication where the source specimen was not available to culture, and the subject was assessed as a clinical cure. To have a favorable microbiological response, the outcome for each participant's baseline pathogen must be favorable (eradicated or presumed eradicated). Other pathogens include Arcanobacterium haemolyticum, Gram positive cocci, Staphylococcus epidermidis, Streptococcus dysgalactiae, Streptococcus mitis group and Streptococcus pyogenes.
Time Frame: Baseline (within 48 hours prior to first dose of IV study drug) - and Test of Cure (21-35 days after last dose of IV study drug) (up to Day 77)
Population: All randomized participants who received IV study drug and had a confirmed diagnosis of AHO, excluding participants with confirmed culture of a gram-negative organism; but including those where at least one bacterial pathogen was isolated from an appropriate microbiological specimen at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 45 | 47
Percentage of participants
  Overall Baseline Infecting Pathogen (n =45,47) | 77.8 [65.6 to 89.9] | 87.2 [77.7 to 96.8]
  Staphylococcus Aureus (SA) (n= 43,42) | 76.7 [64.1 to 89.4] | 88.1 [78.3 to 97.9]
  Methicillin Susceptible SA (MSSA) (n= 39,37) | 79.5 [66.8 to 92.2] | 94.6 [87.3 to 100]
  Methicillin Resistant SA (MRSA) (n= 4,4) | 50.0 [1.0 to 99.0] | 25.0 [0.0 to 67.4]
  Other Pathogens (n= 2,7) | 100 [100 to 100] | 85.7 [59.8 to 100]
Statistical Analysis 1: Comparison: Daptomycin vs Vancomycin or Nafcillin; Overall Baseline Infecting Pathogen; Test type: Superiority or Other; p = 0.230, Wald; Common difference = -10.5, 95% CI 2-sided [-26.3 to 5.4] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Daptomycin vs Vancomycin or Nafcillin; SA; Test type: Superiority or Other; p = 0.164, Wald; Common difference = -12.3, 95% CI 2-sided [-28.5 to 4.4] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Daptomycin vs Vancomycin or Nafcillin; MSSA; Test type: Superiority or Other; p = 0.043, Wald; Common difference = -15.5, 95% CI 2-sided [-31.2 to 1.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Daptomycin vs Vancomycin or Nafcillin; MRSA; Test type: Superiority or Other; p = 0.450, Wald
Statistical Analysis 5: Comparison: Daptomycin vs Vancomycin or Nafcillin; Other Pathogen; Test type: Superiority or Other; p = 0.280, Wald

5. Secondary Outcome: Percentage of Participants With Sustained Clinical Improvement
Description: Sustained clinical improvement was defined as participants with clinical improvement who further met the definition of clinical cure. Clinical improvement was in the three general categories of Pain, Inflammation, and Limb Function on or before Study Day 5. Clinical cure is defined as resolution of all acute symptoms of AHO or improvement to such an extent that no further intravenous antibacterial therapy is required. The EOT visit is within 48 hours of last dose of PO therapy.
Time Frame: Baseline (within 48 hours prior to first dose of IV study drug) - up to Test of Cure (21-35 days after last dose of IV study drug) (up to Day 77)
Population: All randomized participants who received any amount of IV study drug and who had a confirmed or suspected diagnosis of AHO, excluding those with confirmed culture of a gram-negative organism from any baseline specimen; and had non-missing clinical outcome.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 71 | 70
Percentage of participants
  EOT (n= 55,57) | 89.1 [80.9 to 97.3] | 94.7 [88.9 to 100.0]
  TOC (n= 55,58) | 87.3 [78.5 to 96.1] | 91.4 [84.2 to 98.6]
Statistical Analysis 1: Comparison: Daptomycin vs Vancomycin or Nafcillin; EOT; Test type: Superiority or Other; p = 0.272, Wald; Common difference = -6.3, 95% CI 2-sided [-18.2 to 5.5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Daptomycin vs Vancomycin or Nafcillin; TOC; Test type: Superiority or Other; p = 0.480, Wald; Common difference = -4.8, 95% CI 2-sided [-17.6 to 7.9] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response Categorized by Baseline Pathogen at Test of Cure
Description: Favorable microbiological outcomes are either eradication where the source specimen demonstrated absence of the original baseline pathogen; or presumed eradication where the source specimen was not available to culture, and the subject was assessed as a clinical cure. For a favorable microbiological response, the outcome for each baseline pathogen must be eradicated or presumed eradicated. Other pathogens include Arcanobacterium haemolyticum, Gram positive cocci, Staphylococcus epidermidis, Streptococcus dysgalactiae, Streptococcus mitis group and Streptococcus pyogenes.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 45 | 47
Percentage of participants
  Overall Baseline Infecting Pathogen (n =45,47) | 82.2 [71.1 to 93.4] | 91.5 [83.5 to 99.5]
  SA (n= 43,42) | 81.4 [69.8 to 93.0] | 92.9 [85.1 to 100.0]
  MSSA (n= 39,37) | 84.6 [73.3 to 95.9] | 94.6 [87.3 to 100.0]
  MRSA (n= 4,4) | 50.0 [1.0 to 99.0] | 75.0 [32.6 to 100.0]
  Other Pathogens (n= 2,7) | 100 [100.0 to 100.0] | 85.7 [59.8 to 100.0]
Statistical Analysis 1: Comparison: Daptomycin vs Vancomycin or Nafcillin; Overall Baseline Infecting Pathogen; Test type: Superiority or Other; Common difference = -10.1, 95% CI 2-sided [-24.8 to 4.2] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Daptomycin vs Vancomycin or Nafcillin; SA; Test type: Superiority or Other; Common difference = -12.2, 95% CI 2-sided [-27.2 to 2.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Daptomycin vs Vancomycin or Nafcillin; MSSA; Test type: Superiority or Other; Common difference = -10.4, 95% CI 2-sided [-25.4 to 5.2] — [estimate comment as in outcome 2, analysis 1]

7. Other Pre Specified Outcome: Number of Participants With 1 or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, clinically significant laboratory finding, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: Administration of first dose up to approximately six and a half months after last dose of study drug
Population: Treated participants based on the treatment received
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 74 | 72
Participants | 34 | 45

8. Other Pre Specified Outcome: Number of Participants With 1 or More Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that at any dose results in death; is life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or is a congenital anomaly/birth defect.
Time Frame: Administration of first dose through the last follow-up visit; an expected time of up to 6.5 months
Population: Treated participants based on the treatment received
Measure: Number; unit: Participants
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 74 | 72
Participants | 5 | 4

9. Other Pre Specified Outcome: Concentration of Serum Creatine Kinase (CK)
Description: Serum was collected at Baseline and at End of Therapy IV, from which the concentration of CK was determined.
Time Frame: Baseline and End of Therapy IV (up to Day 42)
Population: Treated participants based on the treatment received
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 74 | 72
U/L
  Baseline (n = 68,72) | 141.7 (188.70) | 99.9 (95.00)
  End of Therapy IV (n= 35,41) | 89.4 (66.55) | 82.4 (95.03)

10. Other Pre Specified Outcome: Change From Baseline in Number of Participants With Abnormal Focused (Peripheral) Neurological Assessments
Description: Focused neurological examinations include assessments of alertness, sensation, pupillary reflex and tracking, peripheral reflexes (biceps, patellar tendon, ankle jerk, and plantar response), muscle tone and strength (upper and lower limbs), coordination (finger to nose), and tremor of the hands/fingers.
Time Frame: Baseline and up to Test of Cure (21-35 days after last dose of IV study drug) (up to Day 77)
Population: Data were only summarized for each visit; but not analyzed.
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Plasma Concentration of Daptomycin at the End of IV Infusion
Description: Blood samples were collected, after infusion of IV study drug between the end of infusion on study day 3, up to Day 42
Time Frame: Day 3 up to Day 42
Population: Participants who received a known amount of daptomycin and who had at least one blood sample collected. Participants treated with vancomycin, nafcillin or equivalent were not analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Daptomycin 12 - < 24 Months Old: IV daptomycin 12 mg/kg once daily and ≤3 dummy infusions daily for ages 12 - < 24 months old only.
- Daptomycin 24 Months - < 7 Yrs Old: IV daptomycin 12 mg/kg once daily and ≤3 dummy infusions daily for ages 24 months - < 7 yrs old only.
- Daptomycin 7 - < 12 Yrs Old: IV daptomycin 9 mg/kg once daily and ≤3 dummy infusions daily for ages 7 - < 12 yrs old only.
- Daptomycin 12 - < 18 Yrs Old: IV daptomycin 7 mg/kg once daily and ≤3 dummy infusions daily for ages 12 - < 18 yrs old only.
Arm/Group | Daptomycin 12 - < 24 Months Old | Daptomycin 24 Months - < 7 Yrs Old | Daptomycin 7 - < 12 Yrs Old | Daptomycin 12 - < 18 Yrs Old
Number analyzed (Participants) | 1 | 6 | 5 | 10
µg/mL | 36.800 (0) | 75.772 (39.1156) | 58.940 (27.4149) | 68.907 (56.6695)

12. Other Pre Specified Outcome: Plasma Concentration of Daptomycin at 15 Minutes to 1 Hour After the End of IV Infusion
Description: Blood samples were collected, after infusion of IV study drug between the end of infusion on study day 3, up to Day 42
Time Frame: Day 3 up to Day 42
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Daptomycin 12 - < 24 Months Old | Daptomycin 24 Months - < 7 Yrs Old | Daptomycin 7 - < 12 Yrs Old | Daptomycin 12 - < 18 Yrs Old
Number analyzed (Participants) | 3 | 8 | 12 | 10
µg/mL | 65.533 (30.8468) | 84.564 (35.0179) | 70.342 (35.0196) | 57.370 (61.5616)

13. Other Pre Specified Outcome: Plasma Concentration of Daptomycin at 2 to 3 Hours After the End of IV Infusion
Description: Blood samples were collected, after infusion of IV study drug between the end of infusion on study day 3, up to Day 42
Time Frame: Day 3 up to Day 42
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Daptomycin 7 - < 12 Yrs Old: IV daptomycin 9, mg/kg once daily and ≤3 dummy infusions daily for ages 7 - < 12 yrs old only.
Arm/Group | Daptomycin 12 - < 24 Months Old | Daptomycin 24 Months - < 7 Yrs Old | Daptomycin 7 - < 12 Yrs Old | Daptomycin 12 - < 18 Yrs Old
Number analyzed (Participants) | 0 | 6 | 5 | 9
µg/mL |  | 51.150 (16.1179) | 31.200 (14.7027) | 46.756 (51.2678)

14. Other Pre Specified Outcome: Plasma Concentration of Daptomycin at 4 to 5 Hours After the End of IV Infusion
Description: Blood samples were collected, after infusion of IV study drug between the end of infusion on study day 3, up to Day 42
Time Frame: Day 3 up to Day 42
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Daptomycin 12 - < 24 Months Old | Daptomycin 24 Months - < 7 Yrs Old | Daptomycin 7 - < 12 Yrs Old | Daptomycin 12 - < 18 Yrs Old
Number analyzed (Participants) | 3 | 7 | 11 | 10
µg/mL | 35.933 (6.3956) | 53.059 (21.8879) | 50.809 (26.0469) | 41.447 (57.8657)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (AEs): Up to approximately six and a half months after last dose of study drug. Non-serious AEs (NSAEs): Up to 35 days after last dose of study drug
Description: Treated participants based on the treatment received
Arm/Group | Daptomycin | Vancomycin or Nafcillin
Serious Adverse Events (participants affected / at risk) | 5/74 | 4/72
Other Adverse Events (participants affected / at risk) | 6/74 | 24/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=74) | Vancomycin or Nafcillin (N=72)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=74) | Vancomycin or Nafcillin (N=72)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6)
Pyrexia (General disorders) | 2 (2) | 5 (6)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data generated in this clinical study are the exclusive property of the Sponsor and are confidential. The Sponsor will make all reasonable efforts to publish the results of the study in an appropriate peer-reviewed journal. Authorship on the primary publication of the results from this study will be based on contributions to study design, enrollment, data analysis, and interpretation of results.